CLINICAL TRIAL: NCT06286280
Title: Removal of Cytokines With Cytosorbents After Inflammatory Response Reaction During Cardiac Surgery and Association of Endothelial Progenitor Cells
Brief Title: Removal Of CytoKines With cytoSorbenTs After Inflammatory Response Reaction During Cardiac Surgery
Acronym: ROCKSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Principal Investigator, Zulfugar Timur Taghiyev, Principal Investigator, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AZ221/21; F/23/22 (Other Grant/Funding Number: German Foundation of Heart Research)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Response
Keywords: CD34+ endothelial progenitor cells; systemic inflammation; extracorporeal circulation

STUDY DESIGN:
Intervention Model Description: single-center, two-arm randomized-controlled prospective study
Who Masked: Participant
Masking Description: Participant will not be informed about group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytosorb group (Experimental): Use of hemoadsorber for removal of cytokines. Participants undergoing cardiac surgery will be treated using a hemoadsorption device (CytoSorb) within the cardiopulmonary Bypass circuit (=Intervention)
  Interventions: Device: cytokine adsorber (CytoSorb®)
- Control group (No Intervention): Participants undergoing cardiac surgery will be treated according to Standard of care (no hemoadsorption advice installed in the CPB circuit)

INTERVENTIONS:
Device: cytokine adsorber (CytoSorb®) — binding of cytokines to the sorbent polystyrene of the adsorber during cardiac surgery with extracorporeal circulation
  Arms: Cytosorb group

SUMMARY:
Detailed knowledge about the association between systemic inflammation and endothelial progenitor cell (EPCs) activation during extracorporeal circulation (ECC) is lacking.

This pilot study aims to clarify the relationship between CD34-positive EPCs and cytokine release during ECC using the cytokine adsorber to make a predictive statement regarding the clinical expression of inflammation.

DETAILED DESCRIPTION:
Mechanical cardiovascular support procedures are used as part of cardiac surgery. Here, heart-lung machines (HLM) and miniaturized systems such as ECMO (extracorporeal membrane oxygenation) are used to replace cardiac and/or pulmonary function. Contact with non-physiologic artificial surfaces can induce a generalized 'sterile' inflammatory syndrome called SIRS (Systemic Inflammatory Response Syndrome). During SIRS, proinflammatory cytokine release occurs due to complement activation. These massively released, diverse cytokines significantly influence the activation and release of endothelial progenitor cells (EPCs) from the bone marrow during extracorporeal circulation (ECC) and their long-term functionality.

The life-threatening complications of the so-called cytokine storm can potentially be avoided with the help of a cytokine adsorber (CytoSorb®), and the stabilization process after the hyperinflammatory phase can be promoted. However, it is unclear the quantitative and qualitative modification of the cytokine expression pattern by the use of the cytokine adsorber and its influence on the release of EPCs as well as on the clinical course of the patients. Although a therapy extension with cytokine adsorber has a positive impact on the reduction of cytokine levels in the blood, cytokine removal has not been investigated in direct correlation to EPCs.

These interactions are to be investigated within the scope of the proposed project.

This project is a pilot study with a translational science background to clarify the relationship between CD34-positive endothelial progenitor cells and cytokine release in the setting of ECCs using cytokine adsorber. Previous studies have shown a positive association between increased cytokine levels and the number of circulating endothelial progenitor cells. To date, it has not been investigated how this correlation or association changes with the use of cytokine adsorbers. Therefore, due to the specificity of targeted cytokine removal, the findings obtained here may provide essential insights in basic clinical research that could be applied to clinical issues and decision-making processes in the future. Due to the increasingly important role of extracorporeal circulatory support systems, detailed knowledge of the relationship between systemic inflammation and endothelial progenitor cell activation during their use will be increasingly important in the future.

The current project aims to investigate whether an association between the inflammatory response during and after cardiac surgery and the number of stem cells (EPCs) continues to exist when the cytokine adsorber (CytoSorb®) is applied and whether and how the adsorber can influence the functionality, migratory capacity, and differentiation of stem cells. We assume that under these conditions, a direct correlation of EPCs with inflammation does not exist, so a modulation of the SIRS (Systemic Inflammatory Response Syndrome) clinically observed by us could be absent. In addition, we will investigate whether a correlation between the number of circulating endothelial progenitor cells (CD 34+ cells) and the concentration of cytokines can be observed to make a predictive statement regarding the clinical expression of inflammation.

The long-term goal is to identify patients at high risk for clinical manifestations of inflammation after using the EPC and, based on the knowledge gained, make a predictive statement based on the concentration pattern of the EPC.

This prospective study should provide information on whether and at which point perioperative hyperinflammation can be reliably predicted and whether establishing a specific cytokine adsorber could positively influence the number of EPCs and, thus, short- and medium-term survival.

ELIGIBILITY:
Inclusion Criteria:

* planned cardiac surgical procedure with the use of the cardiopulmonary machine as well as with ECMO use (elective or urgent)
* age at the time of surgery of >18 years.
* informed consent

Exclusion Criteria:

* An emergency indication;
* endocarditis, a non-sterile inflammation,
* autoimmune diseases, chronic inflammatory diseases (ankylosing spondylitis, psoriasis, rheumatoid arthritis, chronic inflammatory intestinal diseases), an acquired immune deficit (HIV);
* severe liver dysfunction, hepatitis B/0;
* patients on dialysis;
* Patients with a hematopoietic disorder/tumour disease;
* participation in other interventional trials or studies;
* timely and probable follow-up cannot be guaranteed (e.g. due to long distances between home and study site); a pregnancy that cannot be excluded with certainty (no menopause, no sterilization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
correlation of endothelial progenitor cells with cytokine levels with and without adsorber use | 24 hours before until day 7 post-surgery
  How does the number of EPCs during adsorber use correlate with cytokine levels, and how does the adsorber influence the time course of EPC release (measurement before and after adsorber use)?

SECONDARY OUTCOMES:
Overall mortality rate | until day 30 post surgery
  Overall mortality rate until day 30
Days on ventilator, vasopressor and renal replacement therapy | until day 30 post-surgery
  Total days on ventilator, vasopressor and renal replacement therapy within 30 days post-surgery will be assessed
incidence of stroke | until day 30 post-surgery
  incidence of stroke within 30 days post-surgery will be assessed
length of ICU and in-hospital stay | until day 30 post-surgery
  total length of ICU and in-hospital stay until day 30 post-surgery
Echocardiographic changes | 24 hours before until day 7 post-surgery
  Does a cytokine adsorber influence left ventricular function?
Influence of Cytokine on endothelial progenitor cells | 24 hours before and immediately after surgery
  Does a cytokine adsorber influence EPC function? After isolation (CD34 sorting) and cultivation in stem cell medium, EPCs will be functionally characterized using angiogenesis assays (sprouting assay; tube formation), migration assays and measurement of DiI-Ac-LDL uptake.

CONTACTS AND LOCATIONS:
Locations (1):
- Universityhospital Giessen, Department of Cardiovascular Surgery, Giessen, Germany, Germany

IPD SHARING:
Plan to Share IPD: Undecided